CLINICAL TRIAL: NCT03992066
Title: A Phase 1b, Randomized, Open-Label Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Vadadustat in Hemodialysis Subjects With Anemia Associated With Chronic Kidney Disease
Brief Title: Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Vadadustat in Hemodialysis Subjects With Anemia Associated With Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0034
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Anemia Associated With Chronic Kidney Disease
Keywords: Anemia; Chronic kidney disease; Vadadustat; Hemodialysis; Erythropoiesis-stimulating agent
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — vadadustat; Darbepoetin alfa; Epoetin Alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Vadadustat 600 mg (Experimental): Dialysis-dependent chronic kidney disease (DD-CKD) participants converting from erythropoiesis-stimulating agent (ESA) treatment will be administered fixed-dose treatment for 10 days with vadadustat 600 milligrams (mg) daily.
  Interventions: Drug: Vadadustat
- Vadadustat 750 mg (Experimental): DD-CKD participants converting from ESA treatment will be administered fixed-dose treatment for 10 days with vadadustat 750 mg daily.
  Interventions: Drug: Vadadustat
- Vadadustat 900 mg (Experimental): DD-CKD participants converting from ESA treatment will be administered fixed-dose treatment for 10 days with vadadustat 900 mg daily.
  Interventions: Drug: Vadadustat
- Erythropoiesis-stimulating agent (Other): Participants will continue to receive their existing treatment with intravenous erythropoiesis-stimulating agent (ESA; darbepoetin alfa or epoetin alfa) for 10 days.
  Interventions: Drug: Darbepoetin alfa; Drug: Epoetin alfa

INTERVENTIONS:
Drug: Vadadustat — oral 150 mg tablet
  Other Names: AKB-6548
  Arms: Vadadustat 600 mg; Vadadustat 750 mg; Vadadustat 900 mg
Drug: Darbepoetin alfa — solution intravenous injection
  Arms: Erythropoiesis-stimulating agent
Drug: Epoetin alfa — solution for intravenous injection
  Arms: Erythropoiesis-stimulating agent

SUMMARY:
This study will be conducted to assess the pharmacokinetics of vadadustat 600, 750, and 900 milligrams daily, and intravenous erythropoiesis-stimulating agent (darbepoetin alfa or epoetin alfa), in hemodialysis participants with anemia associated with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age at the time of informed consent
* Receiving chronic, outpatient in-center hemodialysis three times a week for end-stage renal disease for at least 12 weeks prior to Screening
* Maintained on intravenous erythropoiesis-stimulating agent (ESA) therapy (mean dose of <1.5 micrograms per kilogram per week for darbepoetin alfa, or mean dose of <300 Units per kilogram per week for epoetin alfa) for 8 weeks prior to randomization
* Two hemoglobin values between 8.5 and 10.5 grams per deciliter, inclusive, measured at least 4 days apart within 28 days prior to randomization
* Investigator determines the participant is not likely to need rescue therapy (ESA administration or red blood cell transfusion) or require interruption or discontinuation of study drug within the next 30 days
* Serum ferritin ≥100 nanograms per milliliter and transferrin saturation ≥20% within the 28-day screening period prior to randomization
* Folate and vitamin B12 measurements ≥ lower limit of normal within the 28-day screening period prior to randomization
* Hemodialysis adequacy (Kt/Vurea) as indicated by single-pool Kt/Vurea ≥1.2 using the most recent historical measurement within 12 weeks prior to randomization
* Female participants of childbearing potential who are non-lactating, not pregnant as confirmed by a negative serum pregnancy test at Screening within 9 days prior to dosing on Day 1, and using, and agree to continue using, an acceptable method of contraception for at least 4 weeks prior to first dose of study drug until 30 days after the last dose of study drug. Acceptable contraceptive use is outlined in the protocol.
* Female participants of non-childbearing potential who are either surgically sterile (e.g., hysterectomy, bilateral tubal ligation, bilateral oophorectomy) or post-menopausal (>12 months of spontaneous and continuous amenorrhea in a female >55 years old, or >12 months of spontaneous and continuous amenorrhea with a follicle stimulating hormone [FSH] level >40 International Units per Liter in a female <55 years old)
* Female participants of childbearing potential who agree not to donate ova during the study and for at least 30 days after the last dose of study drug
* Male participants who have not had a vasectomy must agree to use an acceptable method of contraception from time of first dose of study drug until 30 days after the last dose of the study drug, and to not donate sperm during the study and for at least 30 days after the last dose of study drug. Acceptable contraceptive use is outlined in the protocol.
* Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Treated with any HMG-CoA reductase inhibitor (statin) other than atorvastatin, pravastatin, simvastatin, or rosuvastatin within the 28-day screening period prior to randomization. Within the 28-day screening period prior to randomization, the maximum allowable dose of simvastatin is 20 milligrams (mg) daily, and the maximum allowable dose of rosuvastatin is 10 mg daily. These restrictions also apply to the dosing period.
* Treated with clinically relevant substrates of the breast cancer resistant protein (BCRP) transporter (e.g., sulfasalazine, methotrexate, mitoxantrone, imatinib, irinotecan, lapatinib, topotecan, tenofovir, glecaprevir, pibrentasir, or sofosbuvir) within 30 days prior to randomization
* Anemia with a cause other than chronic kidney disease (e.g., sickle cell disease, myelodysplastic syndromes, bone marrow fibrosis, hematologic malignancy, myeloma, hemolytic anemia, thalassemia, or pure red cell aplasia)
* Active bleeding or blood loss within 8 weeks prior to randomization
* Red blood cell transfusion within 8 weeks prior to randomization
* Anticipated to discontinue hemodialysis or change dialysis modality during the study
* History of chronic liver disease (e.g., chronic infectious hepatitis, chronic autoimmune liver disease, cirrhosis or fibrosis of the liver)
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT), or total bilirubin >1.5× upper limit of normal (ULN) within the 28-day screening period prior to randomization. Participants with a history of Gilbert's syndrome may participate in the study if they are not jaundiced, have a total bilirubin <3 × ULN and AST and ALT are not >1.5× ULN.
* Current uncontrolled hypertension that would contraindicate the use of darbepoetin alfa or epoetin alfa as determined by the investigator
* Acute coronary syndrome (hospitalization for unstable angina or myocardial infarction), surgical or percutaneous intervention for coronary, cerebrovascular, or peripheral artery disease (aortic or lower extremity), surgical or percutaneous valvular replacement or repair, sustained ventricular tachycardia, hospitalization for heart failure (HF) or New York Heart Association Class IV HF, or stroke within 12 weeks prior to randomization
* History of new or recurrent malignancy within 2 years prior to Screening or currently receiving treatment or suppressive therapy for cancer. Participants with treated basal cell carcinoma of skin, curatively resected squamous cell carcinoma of skin, or cervical carcinoma in situ may participate on the study.
* History of deep vein thrombosis or pulmonary embolism within 12 weeks prior to randomization
* History of hemosiderosis or hemochromatosis
* History of bilateral native nephrectomy
* History of functioning organ transplantation other than corneal transplant
* Scheduled organ transplant from a living donor or on the kidney transplant wait list or expected to receive a transplant during the study
* History of a prior hematopoietic stem cell or bone marrow transplant (stem cell therapy for knee arthritis is not excluded)
* Known hypersensitivity to vadadustat excipients, or to darbepoetin alfa or epoetin alfa
* Use of an investigational drug within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to randomization
* Prior administration of an hypoxia-inducible factor prolyl-hydroxylase, including vadadustat
* Any other reason, which in the opinion of the investigator, would make the participant not suitable for participation in the study
* Treated with probenecid within the 28-day Screening Period prior to randomization or during the study treatment duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Mean area under concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | Vadadustat: Days 1, 2, 8, and 10 (or End of Treatment). Erythropoiesis-stimulating agent: Days 1 and 2
  Vadadustat: Day 1: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose and prior to dosing. Day 8: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 10 or End of Treatment: predose. Erythropoiesis-stimulating agent: Day 1: predose; 0.25, 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose
Area under concentration-time curve from time 0 to infinity (AUCinf) | Vadadustat: Days 1, 2, 8, and 10 (or End of Treatment). Erythropoiesis-stimulating agent: Days 1 and 2
  Vadadustat: Day 1: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose and prior to dosing. Day 8: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 10 or End of Treatment: predose. Erythropoiesis-stimulating agent: Day 1: predose; 0.25, 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose
Maximum observed concentration (Cmax) | Vadadustat: Days 1, 2, 8, and 10 (or End of Treatment). Erythropoiesis-stimulating agent: Days 1 and 2
  Vadadustat: Day 1: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose and prior to dosing. Day 8: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 10 or End of Treatment: predose. Erythropoiesis-stimulating agent: Day 1: predose; 0.25, 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose
Time to maximum observed concentration (Tmax) | Vadadustat: Days 1, 2, 8, and 10 (or End of Treatment). Erythropoiesis-stimulating agent: Days 1 and 2
  Vadadustat: Day 1: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose and prior to dosing. Day 8: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 10 or End of Treatment: predose. Erythropoiesis-stimulating agent: Day 1: predose; 0.25, 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose
Terminal half-life (t½) | Vadadustat: Days 1, 2, 8, and 10 (or End of Treatment). Erythropoiesis-stimulating agent: Days 1 and 2
  Vadadustat: Day 1: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose and prior to dosing. Day 8: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 10 or End of Treatment: predose. Erythropoiesis-stimulating agent: Day 1: predose; 0.25, 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose
Apparent clearance (CL/F) or clearance (CL) | Vadadustat: Days 1, 2, 8, and 10 (or End of Treatment). Erythropoiesis-stimulating agent: Days 1 and 2
  Vadadustat: Day 1: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose and prior to dosing. Day 8: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 10 or End of Treatment: predose. Erythropoiesis-stimulating agent: Day 1: predose; 0.25, 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose
Apparent volume of distribution (Vd/F) or volume of distribution (Vd) | Vadadustat: Days 1, 2, 8, and 10 (or End of Treatment). Erythropoiesis-stimulating agent: Days 1 and 2
  Vadadustat: Day 1: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose and prior to dosing. Day 8: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 10 or End of Treatment: predose. Erythropoiesis-stimulating agent: Day 1: predose; 0.25, 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose
Tmax for vadadustat metabolite(s) | Day 1: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose and prior to dosing. Day 8: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 10 or End of Treatment: predose
AUClast for vadadustat metabolite(s) | Day 1: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose and prior to dosing. Day 8: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 10 or End of Treatment: predose
AUCinf for vadadustat metabolite(s) | Day 1: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose and prior to dosing. Day 8: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 10 or End of Treatment: predose
Cmax for vadadustat metabolite(s) | Day 1: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose and prior to dosing. Day 8: predose; 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 10 or End of Treatment: predose
Serum erythropoietin concentration for the erythropoiesis-stimulating agent treatment group | Day 1: predose; 0.25, 1, 2, 3, 4, 5, 8, and 11 hours post dose. Day 2: 24 hours (-2 hours) post Day 1 dose

SECONDARY OUTCOMES:
Hepcidin concentration | predose on Days 1, 6, and 10
Serum erythropoietin concentration | predose on Days 1, 6, and 10; post dose on Days 1 and 8
Iron concentration | predose on Days 1, 6, and 10
Ferritin concentration | predose on Days 1, 6, and 10
Total iron-binding capcity | predose on Days 1, 6, and 10
Transferrin saturation | predose on Days 1, 6, and 10
Hemoglobin concentration | post dose on Days 1, 6, and 10
Reticulocyte concentration | predose on Days 1, 6, and 10
Number of participants with any treatment-emergent adverse event | up to Day 40, plus or minus 3 days
Number of participants with clinically significant electrocardiogram findings | up to Day 40, plus or minus 3 days
Number of participants with clinically significant vital sign values | up to Day 40, plus or minus 3 days
Number of participants with clinically significant clinical laboratory values | up to Day 40, plus or minus 3 days

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Research Site, Escondido, California
  - Research Site, Denver, Colorado
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Kansas City, Missouri
  - Research Site, Midwest City, Oklahoma
  - Research Site, Providence, Rhode Island
  - Research Site, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Navarro-Gonzales P, Chavan A, Wang D, Burke SK, Dykstra K. A randomized trial to evaluate the pharmacokinetics, pharmacodynamics, and safety of vadadustat in patients with anemia associated with chronic kidney disease receiving hemodialysis. BMC Nephrol. 2025 Aug 11;26(1):453. doi: 10.1186/s12882-025-04367-x. PMID 40790188
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278